CLINICAL TRIAL: NCT06599502
Title: A Phase I/IIa, Open-label, Multi-centre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AZD0022 Monotherapy and in Combination With Anti-cancer Agents in Participants With Tumours Harbouring a KRASG12D Mutation (ALAFOSS-01)
Brief Title: A Phase I/IIa Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AZD0022 as Monotherapy and in Combination With Anti-cancer Agents in Adult Participants With Tumours Harbouring a KRASG12D Mutation
Acronym: ALAFOSS-01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7080C00001
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumours; Non-Small Cell Lung Cancer (NSCLC); Pancreatic Ductal Adenocarcinoma (PDAC); Colorectal Cancer (CRC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: This protocol has a modular design, with the potential for future Modules or treatment to be added via protocol amendments. Participants will receive oral doses of AZD0022, either as monotherapy or in combination with other anti-cancer agents
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Module 1 Part A. Dose Escalation (Experimental): AZD0022 monotherapy
  Interventions: Drug: AZD0022
- Module 1 Part B. Dose Optimisation (Experimental): AZD0022 monotherapy
  Interventions: Drug: AZD0022
- Module 1 Part C. Potential Efficacy Expansion (Experimental): AZD0022 monotherapy
  Interventions: Drug: AZD0022
- Module 1 Part B. Food Effect Cohort (Experimental): AZD0022 monotherapy
  Interventions: Drug: AZD0022
- Module 2 Part A. Dose Escalation (Experimental): AZD0022 in combination with Cetuximab
  Interventions: Drug: AZD0022; Drug: Cetuximab
- Module 2 Part B. Dose Optimisation (Experimental): AZD0022 in combination with Cetuximab
  Interventions: Drug: AZD0022; Drug: Cetuximab
- Module 2 Part C. Potential Efficacy Expansion (Experimental): AZD0022 in combination with Cetuximab
  Interventions: Drug: AZD0022; Drug: Cetuximab

INTERVENTIONS:
Drug: AZD0022 — AZD0022 is an oral KRASG12D inhibitor that blocks KRASG12D function in patients with this type of mutation.
Drug: Cetuximab — Cetuximab (Erbitux®) is a recombinant chimeric human/mouse Immunoglobulin G monoclonal antibody which binds to EGFR and competitively inhibits the binding of EGFR and other ligands
  Arms: Module 2 Part A. Dose Escalation; Module 2 Part B. Dose Optimisation; Module 2 Part C. Potential Efficacy Expansion

SUMMARY:
This is a first-in-human, modular, Phase I/IIa, open-label, multi-centre study to assess the safety, tolerability, PK, and preliminary efficacy of AZD0022 monotherapy in combination with other anti-cancer agents in participants with tumours harbouring a KRASG12D mutation.

DETAILED DESCRIPTION:
This first time in human, open-label, multi-centre study will administer AZD0022 orally to participants with tumours harbouring a KRASG12D mutation.

This study will have initially 2 modules.

* Module 1: AZD0022 monotherapy
* Module 2: AZD0022 in combination with other anti-cancer agents (Cetuximab)

Each Module has 3 parts. Dose Escalation (Part A), Dose Optimisation (Part B) and Potential Efficacy Expansion (Part C).

ELIGIBILITY:
Key Inclusion Criteria:

For whole study:

1. Participant must be ≥ 18 years or the legal age of consent in the jurisdiction in which the study is taking place at the time of signing the ICF.
2. Participants must have a histologically or cytologically confirmed metastatic or locally advanced tumour. Further details on tumour types are specified in Module-specific inclusion criteria.
3. Participants must have received and progressed on, are refractory or are intolerant to standard therapy for the specific tumour type, or as per Module-specific criteria. Participants with contraindications to, or who refuse SoC therapy may be considered, provided that it is documented and the participant has been informed about all available therapeutic options.
4. Documented KRASG12D mutation in tissue or liquid biopsy.
5. Provision of a FFPE tumour sample.
6. Participants must have at least one measurable target lesion per RECIST v1.1.
7. Adequate organ and marrow function as defined in study protocol.

Module 1 Key Inclusion Criteria

1. Type of tumours with a KRASG12D mutation:

   1. For NSCLC: Patients must have NSCLC that is not amenable to curative treatment and should have progressed on at least one prior line of SoC treatment for metastatic NSCLC (including but not limited to platinum-based chemotherapy, immunotherapy, targeted therapy or first line SoC combinations); prior experimental treatments are allowed.
   2. For CRC: Patients must have CRC that is not amenable to curative treatment and should have progressed on at least 2 prior lines of SoC treatment for metastatic CRC; prior experimental treatments are allowed.
   3. For PDAC: Patients must have PDAC that is not amenable to curative treatment and should have progressed at least one prior line of SoC treatment for metastatic PDAC (including but not limited to FOLFIRINOX, gemcitabine plus abraxane and gemcitabine monotherapy); prior experimental treatments are allowed.
   4. For patients enrolled in Part C (NSCLC and PDAC): at least one but no more than 2 lines of prior treatment in metastatic settings; prior experimental treatments are allowed.
2. Progression or recurrence of the disease within 6 months of completing neo/adjuvant treatment (ie, chemotherapy, immunotherapy, chemoradiotherapy, etc) will be considered as a first line of treatment.
3. For Part B food-effect cohort, participants must be able to eat a standard high-fat meal and must be able to fast for at least 10 hours.

Module 2 Inclusion Criteria

1. For Part A (M2A, dose escalation) participants must have pathologically documented locally advanced or metastatic CRC with a KRASG12D mutation.
2. For Part B (M2B, dose optimisation) participants must have pathologically documented locally advanced or metastatic, PDAC or CRC with a KRASG12D mutation.
3. For Part C (M2C, potential efficacy expansion) participants must have pathologically documented locally advanced or metastatic CRC with a KRASG12D mutation.

4(a) For CRC: Patients must have CRC that is not amenable to curative treatment and should have progressed on at least 2 prior lines of SoC treatment for metastatic CRC; prior treatment are allowed.

(b) For PDAC: Patients must have PDAC that is not amenable to curative treatment and should have progressed at least one prior line of SoC treatment for metastatic PDAC (including but not limited to FOLFIRINOX, gemcitabine plus abraxane and gemcitabine monotherapy); prior experimental treatment are allowed.

(c) For patients enrolled in Part C (M2C), at least 2 but no more than 3 lines of prior treatment in metastatic setting; prior experimental treatment are allowed.

5. Progression or recurrence of the disease within 6 months of completing neo/adjuvant treatment (ie, chemotherapy, immunotherapy, and chemoradiotherapy) will be considered as a first line of treatment.

Exclusion Criteria:

For whole study:

1. Any significant laboratory finding or any severe and uncontrolled medical condition.
2. Any evidence of clinically significant current or prior ILD (eg, required IV steroids or high supplemental oxygen) or where a new suspected ILD cannot be ruled out by imaging at screening.
3. Spinal cord compression, leptomeningeal disease, or active brain metastases. Asymptomatic brain metastases are allowed
4. History of allogenic organ transplantation.
5. Participants with any of the following cardiac criteria:

   * Mean resting QTcF > 470 milliseconds on screening
   * Any factors that increase the risk of QT prolongation
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, second- or third-degree atrioventricular block), and clinically significant sinus node dysfunction not treated with pacemaker.
   * Bradycardia defined as a heart rate less than 60 beats per minute and/or hypotension defined as a blood pressure reading lower than 90 mm Hg for the top number (systolic) or 60 mm Hg for the bottom number (diastolic).
   * Baseline LVEF below the institutional lower limit of normal or < 50%, whichever is lower.
   * Symptomatic heart failure (as defined by New York Heart Association class ≥ 2).
   * Acute coronary syndrome/acute myocardial infarction, unstable angina pectoris, coronary intervention procedure with percutaneous coronary intervention, or coronary artery bypass grafting within 6 months before C1D1.
6. Prior exposure to any direct small molecule KRAS inhibitor.
7. Herbal preparations/medications are not allowed during treatment with study drug.
8. Any concomitant medications that are known strong inhibitors or inducers of CYP3A4/5, or sensitive CYP3A4/5 substrates or CYP3A4/5 substrates with a narrow therapeutic range. This also applies to moderate inhibitors and moderate inducers of CYP3A4/5 during Parts A and B of Modules 1 and 2.
9. Receipt of a cytotoxic or non-cytotoxic drug: 21 days or 5 half-lives, whichever is shorter, before the first dose of study intervention. Biological therapy including immune-oncology and monoclonal antibodies 28 days or 5 half-lives.
10. Less than or equal to 4 weeks for radiation therapy given with curative intent or ≤ 2 weeks for limited field radiation for palliation prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with Dose-Limiting Toxicity (DLT), Adverse events (AEs) and Serious Adverse Events (SAEs). | From time of informed consent, through study completion to 30 days post last dose; an average of 2 years
  Determine if treatment with AZD0022 as a monotherapy and in combination with other anti-cancer agents is safe and tolerable through the assessment of DLTs, AEs, SAEs, and change from baseline in laboratory parameters, vital signs, and ECGs.
  Part A (Dose Escalation) and Part B (Dose Optimisation). DLTs only applicable for Part A.
Number of patients who discontinue AZD0022 due to toxicity | From time of informed consent to 30 days post last dose
  To investigate the safety and tolerability of AZD0022 as a monotherapy and in combination with other anti-cancer agents in participants with advanced tumours harbouring a KRASG12D mutation
  Part A (Dose Escalation) and Part B (Dose Optimisation)
ORR (Objective Response Rate) | Time from first dose of AZD002 through study completion; approximate duration of 2 years
  Evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part C (Potential Efficacy Expansion)
  Percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
CR rate (Complete Response) | From first dose (non-randomised study parts) or from randomisation (randomised) through study completion; approximate duration of 2 years
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion)
  Percentage of participants with a confirmed Complete Response (CR)
DoR (Duration of Response) | From the date of first response until date of disease progression (RECIST 1.1) or death in the absence of disease progression; approximate duration of 2 years.
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion).
  Time from the date of first documented evidence of CR or PR until date of first documented disease progression or death.
DCR (Disease Control Rate) | From first dose (non-randomised study parts) or from randomisation (randomised) until progression. For each patient, this is expected to be at 12 weeks
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion).
  Percentage of participants who have a confirmed CR, PR, or Stable Disease (SD) for at least 11 weeks after start of treatment.
DRR (Durable Response Rate) | From first documented response up until progression, or the last evaluable assessment in the absence of progression; approximate duration of 2 years.
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion).
  Percentage of participants who have a confirmed response (CR/PR) with a duration of at least 3 months.
TTR (Time to Response) | From first dose (non-randomised study parts) or from randomisation (randomised study parts) until the date of documented objective response; approximate duration of 2 years.
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion)
  Time from first dose/randomisation date until date of first documented evidence of CR or PR per RECIST v1.1
PFS (Progression Free Survival) | 'From first dose (non-randomised study parts) or from randomisation (randomised study parts) to progressive disease or death in the absence of disease progression; approximate duration of 2 years
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion).
  Time from first dose/randomisation date until date of first documented disease progression or death.
Change in tumour size | From the first dose of study intervention (non-randomised study parts) or from randomisation (randomised), at predefined intervals throughout the administration of AZD0022; approximate duration of 2 years.
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion)
  Percentage change in tumor size from baseline per RECIST v1.1
OS (Overall Survival) | From first dose of study intervention (non-randomised study parts) or from randomisation (randomised study parts) to death; approximate duration of 2 years.
  To assess the preliminary anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion).
  Time from first dose/randomisation date until death due to any case.
Complete Molecular Response (cMR). | From the first dose of study intervention (non-randomised study parts) or from randomisation (randomised study parts), at predefined intervals throughout the administration of AZD0022; approximate duration of 2 years.
  To assess the molecular response rate via ctDNA on treatment with AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Part A (Dose Escalation), Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion).
Pharmacokinetics of AZD0022: Maximum plasma concentration of the study drug (Cmax) | From the first dose of study intervention (non-randomised study parts) or from randomisation (randomised study parts), at predefined intervals throughout the administration of AZD0022; approximate duration of 2 years.
  Maximum observed plasma concentration of the study drug
  Part A (Dose Escalation) and Part B (Dose Optimisation)
Pharmacokinetics of AZD0022: Time to maximum plasma concentration of the study drug (T-max) | From the first dose of study intervention (non-randomised study parts) or from randomisation (randomised study parts), at predefined intervals throughout the administration of AZD0022; approximate duration of 2 years.
  Time to maximum observed plasma concentration of the study drug
  Part A (Dose Escalation) and Part B (Dose Optimisation)
Pharmacokinetics of AZD0022: AuClast (Area Under the Plasma Contentration-Time Curve to the Last Measurable Plasma Concentration) | From the first dose of study intervention (non-randomised study parts) or from randomisation (randomised study parts), at predefined intervals throughout the administration of AZD0022 until Cycle 3 Day 1.
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time.
  Part A (Dose Escalation) and Part B (Dose Optimisation)
Pharmacokinetics of AZD0022: Terminal elimination half-life (t 1/2) | From the first dose of study intervention (non-randomised study parts) or from randomisation (randomised study parts), at predefined intervals throughout the administration of AZD0022 until Cycle 3 Day 1.
  Terminal elimination half life.
  Part A (Dose Escalation) and Part B (Dose Optimisation)
Incidence of participants with Adverse events (AEs) and Serious Adverse Events (SAEs). | From time of informed consent, through study completion to 30 days post last dose; an average of 2 years
  Determine if treatment with AZD0022 as a monotherapy and in combination with other anticancer agents is safe and tolerable through the assessment of AEs, SAEs, and change from baseline in laboratory parameters, vital signs, and ECGs.
  Part C (Potential Efficacy Expansion).
Number of patients who discontinue AZD0022 due to toxicity | From time of informed consent, through study completion to 30 days post last dose; an average of 2 years
  To further assess the safety and tolerability of AZD0022 as a monotherapy and in combination with other anti-cancer agents
  Part C (Potential Efficacy Expansion).
TDT (Time to Discontinuation of Treatment) | From first dose until discontinuation of treatment for any reason; approximate duration of 2 years.
  To estimate the anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents.
  Part C (Potential Efficacy Expansion)
  Time from first dose/randomisation date until discontinuation of treatment or death due to any case.
TFST (Time to First Subsequent Anti-Cancer) | From date of first dose until start date of the first subsequent anti-cancer therapy after discontinuation of study treatment, or death; approximate duration of 2 years.
  To estimate the anti-tumour activity of AZD0022 as a monotherapy and in combination with other anti-cancer agents.
  Part C (Potential Efficacy Expansion).
  Time from first dose/randomisation date until start of first subsequent anti-cancer therapy after discontinuation of study treatment, or death due to any cause.
Change in phospho-ERK | From baseline, at predefined intervals throughout the administration of AZD0022; approximate duration of 2 years.
  To assess KRAS pathway inhibition on treatment with AZD0022 as monotherapy
  Module 1 Part A (Dose Escalation), Module 1 Part B (Dose Optimisation) and Module 1 Part C (Potential Efficacy Expansion)*
  Module 2 Part A (Dose Escalation), Module 2 Part B (Dose Optimisation) and Module 2 Part C (Potential efficacy expansion)*
  *Potential Efficacy Expansion at Sponsor discretion based on emerging data.
Geometric mean and 90% CI for the ratio of fed:fasted in AUClast and Cmax for food-effect cohort. | From first dose, at predefined intervals throughout the administration of AZD0022; approximate duration of 2 years.
  To characterise the effect of food on AZD0022 as monotherapy
  Module 1 Food-effect only
PFS (Progression Free Survival) by BICR | From first dose (non-randomised study parts) or from randomisation (randomised study parts) to progressive disease or death in the absence of disease progression; approximate duration of 2 years
  To assess anti-tumour activity of AZD0022 as monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Module 1 Part B (Dose Optimisation) and Module 1 Part C (Potential Efficacy Expansion)
  Module 2 Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion)
ORR (Objective Response Rate) by BICR | From first dose (non-randomised study parts) or from randomisation (randomised) through study completion; approximate duration of 2 years
  To assess anti-tumour activity of AZD0022 as monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Module 1 Part B (Dose Optimisation) and Module 1 Part C (Potential Efficacy Expansion)
  Module 2 Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion)
DoR (Duration of Rate) by BICR | From the date of first response until date of disease progression (RECIST 1.1) or death in the absence of disease progression; approximate duration of 2 years.
  To assess anti-tumour activity of AZD0022 as monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Module 1 Part B (Dose Optimisation) and Module 1 Part C (Potential Efficacy Expansion)
  Module 2 Part B (Dose Optimisation) and Part C (Potential Efficacy Expansion)
ORR (Objective Response Rate) by Investigator | From first dose (non-randomised study parts) or from randomisation (randomised) through study completion; approximate duration of 2 years
  To assess anti-tumour activity of AZD0022 as monotherapy and in combination with other anti-cancer agents
  Radiological response evaluated according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours Version 1.1)
  Module 1 Part A (Dose Escalation) and Module 1 Part B (Dose Optimisation)
  Module 2 Part A (Dose Escalation) and Module 2 Part B (Dose Optimisation)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Research Site, Duarte, California
  - Research Site, New York, New York
  - Research Site, Fairfax, Virginia
- Research Site, Melbourne, Australia
- Research Site, Tokyo, Japan
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/